CLINICAL TRIAL: NCT06979817
Title: TLS-Informed Machine Learning Model Predicts Survival and Immune Landscape in Locally Advanced Gastric Cancer
Brief Title: Machine Learning Model Guided by TLS Predicts Survival and Immune Features in Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Qun Zhao (Other)
Responsible Party: Sponsor-Investigator, Qun Zhao, Professor, Hebei Medical University
Organization: Hebei Medical University (Other)
Other Study IDs: GC-RAD-AI-2025-03
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Gastric Cancer; Tumor Immune Microenvironment; Tertiary Lymphoid Structures (TLS)
MeSH Terms: conditions — Tertiary Lymphoid Structures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Locally Advanced Gastric Cancer Patients
  Interventions: Other: TLS-Informed Machine Learning Prognostic Model

INTERVENTIONS:
Other: TLS-Informed Machine Learning Prognostic Model — This intervention involves the development and application of a machine learning-based prognostic model that integrates features derived from tertiary lymphoid structures (TLSs) identified in tumor pathology slides, along with clinical and immunological data, to predict overall survival and immune landscape in patients with locally advanced gastric cancer. The model utilizes digital pathology, image analysis, and advanced computational algorithms to quantify TLS-related characteristics and correlate them with patient outcomes. It is designed to stratify patients into risk groups and provide insight into the tumor immune microenvironment, aiming to support personalized treatment planning.

SUMMARY:
This study aims to develop and validate a machine learning model that uses information from tertiary lymphoid structures (TLSs)-specialized immune-related cell clusters found near tumors-to predict survival outcomes and immune characteristics in patients with locally advanced gastric cancer. By analyzing clinical data, pathology, and imaging results, the model may help doctors better understand a patient's prognosis and personalize treatment strategies. The study will also explore how TLS-related immune patterns relate to the effectiveness of certain therapies, potentially offering new insights for immune-based treatment planning.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed locally advanced gastric adenocarcinoma (clinical stage cT2-T4 and/or N+)

Underwent curative-intent gastrectomy (with or without neoadjuvant therapy)

Availability of adequate tumor tissue specimens for TLS assessment via digital pathology

Complete baseline clinical, pathological, and follow-up data

Age ≥ 18 years

Written informed consent provided (if prospective study component is included)

Exclusion Criteria:

Distant metastases at the time of diagnosis or surgery (M1 stage)

Prior history of other malignancies within the past 5 years, except for adequately treated in situ carcinoma or non-melanoma skin cancer

Incomplete or missing essential clinical, pathological, or survival data

Poor-quality tissue samples not suitable for TLS quantification or digital analysis

Participation in another clinical trial that may interfere with the study outcomes

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will include patients with histologically confirmed locally advanced gastric adenocarcinoma who have undergone curative-intent surgical resection at participating medical centers. The population will consist of both retrospective and prospective cohorts, with all patients having available tumor tissue for TLS analysis and complete clinical, pathological, and follow-up data. The study aims to capture a representative sample of real-world gastric cancer patients, reflecting a diversity of clinical characteristics, treatment modalities, and outcomes.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival Predicted by TLS-Informed Machine Learning Model | Up to 5 Years Post-Surgery